CLINICAL TRIAL: NCT01421212
Title: Study to Assess the Pharmacokinetics of Intravenous Nabi 5% Hepatitis B Immune Globulin Used in Combination With Lamivudine
Brief Title: Pilot Study to Assess the Pharmacokinetics of Intravenous Nabi 5% Hepatitis B Immune Globulin (Boca HBVIg) Used in Combination With Lamivudine for Patients With Hepatitis B Virus (HBV) Associated Liver Disease Undergoing Liver Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotest Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Nabi-4204
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2011-08

CONDITIONS: Hepatitis B Virus Associated Liver Disease
Keywords: Liver Transplantation; Liver Disease; Hepatitis B; Hepatitis B Infection; Hepatitis B Associated Liver Disease; HBV
MeSH Terms: conditions — Liver Diseases; Hepatitis B | interventions — hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Hepatitis B Immune Globulin (Boca HBVIg) — Phase I (12 weeks): Intravenous Boca HBVIg 10,000 IU administered intraoperatively during the anhepatic phase, following reperfusion, daily on days 1-7, once during week 4 and once during week 8 (total of 11 doses).
  Phase II (24 weeks): Starting at 12 weeks post liver transplantation, Boca HBVIg will be reduced to 5,000 IU given intravenously on a monthly basis for patients who had an anti-HBs trough titer greater than or equal to 500 IU/L at 8 weeks without the need for additional Boca HBVIg doses. Patients with an 8 week trough level less than 500 IU/L will receive 10,000 IU Boca HBVIg every 4 weeks for the remainder of the study.
  Other Names: Nabi-HB; HepaGam B; Hepatitis B Immune Globulin; HBIG

SUMMARY:
The purpose of this study is to find the best monthly dose schedule for the new Hepatitis Immune Globulin (Boca HBVIg, a study drug) when used in combination with an antiviral agent Lamivudine after liver transplantation. Boca HBVIg will be given along with Lamivudine to prevent hepatitis B reinfection following liver transplantation in patients with end stage liver failure due to hepatitis B infection.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old or greater, either male or female, of any ethnic background.
* Be positive for HBsAg. Patients may be either positive or negative for anti-HDV, HBeAg, and HBV DNA (non-PCR assay).
* Be diagnosed with HBV-induced liver disease including either:
* HBsAg positive cirrhosis, or
* HBsAg positive and presence of hepatocellular carcinoma (HCC) with no evidence of vascular invasion or extrahepatic spread, and either:
* a single tumor no larger than 5 cm in diameter, or
* no more than three tumors, the largest of which is no greater than 3 cm in diameter.
* Have received at least one dose of Lamivudine 100 mgs po qd prior to transplantation.
* Fulfill UNOS minimal listing criteria.
* Have received approval for liver transplantation at the respective participating center and are listed as Status 2 or 3 and felt to be within three months of liver transplantation.
* If requiring retransplantation for primary graft nonfunction or hepatic artery thrombosis, retransplantation must take place within the first four weeks of the initial transplant with no evidence of recurrent hepatitis B.
* Be able and willing to give written informed consent. In patients with Grade 3 or 4 hepatic encephalopathy, a legal guardian must be available to provide consent. In the case of a minor, a parent or guardian must provide consent.
* If a woman of childbearing potential, have a negative serum beta HCG pregnancy test within 14 days prior to starting Lamivudine therapy and within 14 days prior to transplant and agree to practice contraception during the study (a total of 36 weeks).

Exclusion Criteria:

* Eligible patients must not:
* Require retransplantation for recurrent hepatitis B.
* Have chronic hepatitis B liver disease with a history of breakthrough infection on Lamivudine
* Have other causes of liver disease including chronic hepatitis C.
* Have HCC and do not meet Inclusion Criterion #3, or who require systemic chemotherapy.
* Be seropositive for HIV infection.
* Be using experimental devices or receiving experimental drugs.
* Be participating in any other clinical treatment trial with an investigational drug within 30 days prior to liver transplantation or plan to receive another investigational drug during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-11; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Number of hepatitis B virus positive liver transplant recipients with no hepatitis B virus recurrence after liver transplantation.
Number of participants who maintain a protective trough titer of anti hepatitis B antibodies beginning at 12 weeks post liver transplantation.

SECONDARY OUTCOMES:
Change in anti hepatitis B antibodies levels with administration of Boca hepatitis B immune globulin concomitantly with Lamivudine.

CONTACTS AND LOCATIONS:
Overall Officials: Rolland C. Dickson, M.D., Principal Investigator — Mayo Clinic; Norah A. Terrault, M.D., MPH, Principal Investigator — University of California, San Francisco, CA; Donald Jensen, M.D., Principal Investigator — Rush-Presbyterian - St. Luke's Medical Center, Chicago, IL; Terence Angtuaco, M.D., Principal Investigator — Rush-Presbyterian - St. Luke's Medical Center, Chicago, IL; Patricia Sheiner, M.D., Principal Investigator — Mount Sinai Medical Center, New York, NY; Velimir A. Luketic, M.D., Principal Investigator — Virginia Commonwealth University, Richmond, VA; Michael Fried, M.D., Principal Investigator — University of North Carolina, Chapel Hill, NC; Robert S. Brown, M.D., MPH, Principal Investigator — Columbia-Presbyterian Medical Center, New York, NY; Michael Ishitani, M.D., Principal Investigator — Rochester Methodist Hospital, Rochester, MN; Consuelo Soldevila-Pico, M.D., Principal Investigator — University of Florida; Anna Lok, M.D., Principal Investigator — University of Michigan, Ann Arbor, MI; Rajender Reddy, M.D., Principal Investigator — University of Miami, Miami, FL
Locations (11):
- United States (11):
  - University of California, San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Jackson Memorial Hospital / University of Miami, Miami, Florida
  - Rush-Presbyterian - St. Luke's Medical Center, Chicago, Illinois
  - The University of Michigan Health System, Ann Arbor, Michigan
  - Rochester Methodist Hospital, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - New York-Presbyterian Hospital Columbia-Presbyterian Medical Center, New York, New York
  - The University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Medical College of Virginia Commenwealth University, Richmond, Virginia